CLINICAL TRIAL: NCT05280119
Title: Assessment of the echOpen Ultra-portable Ultrasound Device in Daily Use by Clinicians. Part I: Identification of Effusion and Detection of Basilic Vein
Brief Title: Efficacy of the echOpen Device to Identify Effusion and to Detect Basilic Vein
Acronym: CLIN-ECHO-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: ECHOPEN (Industry); EIT Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: APHP210065; 2021-A00341-40 (Other: IDRCB)
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Pleural Effusion; Abdominal Effusion; Procedural Guidance
Keywords: Ultrasound; Ultrasonography; Point-of-care-ultrasound; Pleural Effusion; Abdominal Effusion; Basilic vein
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Intervention Model Description: A single group, comparative, non-randomized, controlled study. Each patient represents her/his own control: the patient is examined consecutively with the echOpen probe, then with the probe used in the department
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients benefitting ultrasound examination (Experimental): This is the only arm of the study. Patients with an indicative clinical picture that leads the clinician to resort to the use of an ultrasound to potentially support the diagnosis will be examined to verify the presence of pleural effusion or intra-abdominal effusion, or to identify basilic vein. The patients will be assessed first with the echOpen device and second witn an ultrasound routinely used in the department. In a case of discordance between the assessments made with echOpen and the usual ultrasound device, an independent referent radiologist will use a standard ultrasound machine to constitute the gold standard (GS) rating
  Interventions: Device: EchOpen ultra-portable ultrasound device; Device: Ultrasound device routinely used in the department.; Procedure: Standard ultrasound examination by an independent referent radiologist

INTERVENTIONS:
Device: EchOpen ultra-portable ultrasound device — Depending on the clinical picture, patients are examined to detect the presence or absence of pleural effusion, or intra-abdominal effusion, or to localize the basilic vein
Device: Ultrasound device routinely used in the department. — Patients who were first examined with the EchOpen ultra-portable ultrasound device, are secondarily examined with an ultrasound probe used routinely in the department.
Procedure: Standard ultrasound examination by an independent referent radiologist — In a case of discordance between the assessments made with echOpen and the usual ultrasound device, an independent referent radiologist will use a standard ultrasound machine to constitute the gold standard (GS) rating

SUMMARY:
In recent years, portable and ultra-portable ultrasound devices are increasingly used by the non radiologists, notably cardiologists or obstetrician gynecologist, at the patient's bedside to visualize and measure anatomical structures and fluid and provide the clinical examination with additional signs allowing quicker and more confident clinical decisions.

This innovative approach is slowed down by the accessibility of these miniaturized devices, the price of which remains high.

The echOpen device includes an ultra-portable ultrasound probe and a mobile application that allows the image to be displayed on a smartphone via a WIFI protocol.

The objective of the clinical investigation is to show that the echOpen device, using three frequencies 3.5 Mhz, 5.0 Mhz and 7.5 Mhz, allows identifying the semiological signs or anatomical structures of interest located at several depths of the body, with a performance similar to other devices routinely used in clinical departments.

DETAILED DESCRIPTION:
The echOpen device includes an ultrasound probe and a mobile application. The mechanical probe emits at three ultrasound frequencies, 3.5 Mhz, 5.0 Mhz and 7.5 Mhz, which allows the exploration of the interior of the body at different depths in a non-invasive and non-irradiating manner.

Thus, the purpose of the echOpen device is, on one hand, to guide the diagnosis during the clinical examination and, on the other hand, to identify anatomical structures in order to assist in management.

The objective of the clinical investigation is to demonstrate that the echOpen device is able to identify semiological signs and localize anatomical structures at different depths of the body, with a performance not inferior to that of other ultrasound devices, routinely employed in hospital clinical departments.

The signs of interest (i.e. search for an intra-abdominal (3.5 Mhz) and pleural (5.0 Mhz) effusion) were chosen for their clinical usefulness (their presence during the clinical examination constitutes an argument for orientation and/or severity) and for their prevalence in the study population.

The identification of anatomical structure of interest (i.e. detection of basilic vein (7.5Mhz)) was chosen because it is a gesture frequently used when taking in charge of a patient hospitalized in the selected departments.

An ultrasound probe in use in the hospital clinical departments where the investigation takes place will be employed as a comparator to judge the performance of the echOpen device.

This clinical investigation is part of a CE marking procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (age ≥ 18 years old)
* Patient having signed the informed consent to participate in this clinical investigation
* Patient affiliated to the social security scheme
* Patient arriving in the hospital clinical ward (own initiative or by emergency services) whose clinical symptomatology (e.g. dyspnea, thoracic pain, etc.) suggests the presence of pathological elements (effusion) which would be visible using an ultrasound probe
* Patient consulting in the hospital clinical ward who could potentially benefit from a basilic vein line placement using an ultrasound device

Exclusion Criteria:

* Minor patient (age < 18 years)
* Patients under the "State medical assistance"
* Obese patient (body mass index > 29.9)
* Patient in too serious condition for the clinical examination to be done fully and/or with additional exploratory time
* Unstable patient: need for immediate care, impossibility to carry out a thorough clinical examination including interview, palpation, auscultation, percussion
* Known allergy to ultrasound gel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Presence of Pleural effusion | Day 0
  Presence or absence of pleural effusion as assessed by the echOpen device or by a portable ultrasound routinely used in the department
Presence of Intra-abdominal effusion | Day 0
  Presence or absence of intra-abdominal effusion as assessed by the echOpen device or by a portable ultrasound routinely used in the department
Basilic vein identification | Day 0
  Successful identification of the basilic vein using the echOpen device or a portable ultrasound routinely used in the department

SECONDARY OUTCOMES:
Plural effusion detected using a gold standard procedure | Day 0
  Presence of pleural effusion determined by an independent referent radiologist using a standard ultrasound machine
Intra-abdominal effusion detected using a gold standard procedure | Day 0
  Presence or absence of intra-abdominal effusion determined by an independent referent radiologist using a standard ultrasound machine
Basilic vein identification using a gold standard procedure | Day 0
  Identification of the basilic vein by an independent referent radiologist using a standard ultrasound machine

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme BOKOBZA, MD, Principal Investigator — AP-HP, Cochin Hospital
Locations (4):
- France (4):
  - Avicenne Hospital - APHP - Hepatology Department, Bobigny
  - Cochin Hospital - APHP - Emergency Department, Paris
  - Cochin Hospital - APHP - Pneumology department, Paris
  - Paul Brousse Hospital - APHP - Hepatobiliary Center, Villejuif